CLINICAL TRIAL: NCT05502770
Title: Development of IVF/ICSI Children Born From Frozen Embryo Transfer Cycles With Different Endometrial Preparation Protocols: Follow-up of a Randomized Controlled Trial
Brief Title: Development of IVF/ICSI Children Born From Different Endometrial Preparation Protocols
Acronym: MONARTBABIES
Status: Recruiting | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 09/22/DD-BVMD
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Child Development; Endometrial Preparation
Keywords: Child development; Endometrial preparation; IVF/ICSI; Natural cycle; Modified natural cycle; Artificial cycle
MeSH Terms: interventions — Health Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Natural cycle children: Children born from frozen embryo transfer with natural cycle protocol
  Interventions: Diagnostic Test: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Diagnostic Test: Developmental Red flags
- Modified natural cycle children: Children born from frozen embryo transfer with modified natural cycle protocol
  Interventions: Diagnostic Test: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Diagnostic Test: Developmental Red flags
- Artificial cycle children: Children born from frozen embryo transfer with artificial cycle protocol
  Interventions: Diagnostic Test: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Diagnostic Test: Developmental Red flags

INTERVENTIONS:
Diagnostic Test: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3 — Ages & Stages Questionnaires®, Third Edition (ASQ®-3) is a developmental screening tool designed for use by early educators and health care professionals. It relies on parents as experts, is easy-to-use, family-friendly and creates the snapshot needed to catch delays and celebrate milestones.
Other: Physical development and General Health — Physical development and General health examination
Diagnostic Test: Developmental Red flags — Developmental Red flags Questionnaires

SUMMARY:
The efficacy and safety of endometrial preparation regimens remain controversial. In the most recent meta-analysis, using natural and modified natural cycle protocol to prepare the endometrium in frozen embryo transfer resulted in higher live birth rates. In addition, the natural cycle reduces the risk of gestational hypertension, postpartum haemorrhage, and extremely preterm delivery compared with regimens using exogenous hormones.

Because there are many physiological and endocrinal differences in the frozen embryo transfer cycle with different endometrial preparation protocols, the development of children born from these regimens has received much attention. For example, there is a complete absence of the corpus luteum during the cycle of exogenous hormone administration. Or in the modified natural cycle, the pharmacokinetics is not entirely the same as the natural physiology when using an additional ovulatory injection with hCG. To date, there have been no longitudinal follow-up studies that evaluated and compared the long-term development of IVF/ICSI children born from frozen embryo transfer with different endometrial preparation protocols.

Thus, the investigators conduct a follow-up of our RCT to investigate the IVF/ICSI children born from frozen embryo transfer with different endometrial preparation protocols to give strong evidence about the safety of the three most common endometrial preparation protocols in women undergoing frozen embryo transfer.

DETAILED DESCRIPTION:
Developing further from a previous randomized controlled clinical trial (MONART study - NCT04804020), the investigators decided to assess the physical, mental, and motor development of children up to 24 months after birth, with the aim of providing additional information on the safety of these regimens on the long-term health of the IVF/ICSI children.

ELIGIBILITY:
Inclusion Criteria:

* All live IVF/ICSI babies born from frozen embryo transfer following the natural cycle, modified natural cycle, and artificial cycle from MONART study
* Parents agree to participate in the study.

Exclusion Criteria:

* Babies died under or at 24 months

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Live IVF/ICSI babies born from frozen embryo transfer following the natural cycle, modified natural cycle, and artificial cycle from MONART study (NCT04804020)
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The average total ASQ-3 score | Up to 24 months after birth
  ASQ-3 (Ages and Stages Questionaires®) has 5 aspects: Communication, Gross motor, Fine motor, Problem solving and Personal-Social Each aspect has 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  ASQ-3 average = average score of 5 aspects.

SECONDARY OUTCOMES:
Score of Communication | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Gross motor | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Fine motor | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Problem solving | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Personal-Social | Up to 24 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
The rate of children who have at least one red flag sign | From 6 months to 24 months after birth
  He or she has at least one red flag sign by age. For children at 6 months: he or she Lack of turning toward voices. Does not pass object from one hand to another. No smiling, laughing, or expression.
  For children at 12 months: he or she Child does not respond to name. Does not understand "no". Does not stand or bear weight on legs when supported. Indifferent or resistant attachment to caregiver. Does not look where caregiver points.
  For children at 18 months: he or she has Not using at least 6 words. Inability to walk independently. Absence of proto-imperative pointing (point to show interest) or showing gesture.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, Study Chair — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam